CLINICAL TRIAL: NCT06491355
Title: Efficacy and Safety of First-Line Treatment Induced With mFOLFOX6 and HLX04 Regimen, Following Combined With Serplulimab in MSS Initially Unresectable Metastatic Colorectal Cancer: A Prospective, Multicenter, Randomized, Controlled Trial (ASTRUM-IUmCRC)
Brief Title: First-Line Treatment Induced With mFOLFOX6 and HLX04 Regimen, Following Combined With Serplulimab in MSS Initially Unresectable Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Zhangfa Song, Professor, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASTRUM-IUmCRC
Record Dates: First submitted 2024-06-25; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Efficacy, Self; Safety Issues; Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mfolfox6 and hlx04 regimen induction therapy followed by combined treatment with slulimumab (Experimental): Induction therapy: mFOLFOX6 regimen + bevacizumab. lasting 2 cycles. Combination therapy: mFOLFOX6 regimen + bevacizumab + PD-1 monoclonal antibody. Every 2 weeks is a cycle.
  Interventions: Drug: mfolfox6 and hlx04 regimen and Serplulimab
- mfolfox6 and hlx04 regimen treatment (Active Comparator): mFOLFOX6+ HLX04 (bevacizumab). The mFOLFOX6 regimen is: oxaliplatin, calcium leucovorin, 5-fluorouracil, bevacizumab, One cycle is every 2 weeks, lasting 2 cycles.
  During treatment, the drug was administered continuously, and tumor response was assessed by imaging every 8 weeks.
  Interventions: Drug: mfolfox6 and hlx04 regimen

INTERVENTIONS:
Drug: mfolfox6 and hlx04 regimen and Serplulimab — mfolfox6 and hlx04 regimen induction therapy followed by combined treatment with slulimumab in the experimental arm. In the active comparator. only with mfolfox6 and hlx04 regimen treatment.
  Arms: mfolfox6 and hlx04 regimen induction therapy followed by combined treatment with slulimumab
Drug: mfolfox6 and hlx04 regimen — In the active comparator. only with mfolfox6 and hlx04 regimen treatment.
  Arms: mfolfox6 and hlx04 regimen treatment

SUMMARY:
This is a prospective, multi-center, randomized controlled clinical intervention study, aiming to explore the effectiveness and safety of mfolfox6 and hlx04 regimens combined with slulimumab as first-line treatment for MSS-type initial unresectable metastatic colorectal cancer after induction therapy. This study plans to include a total of 72 patients with untreated MSS-type initial unresectable metastatic colorectal cancer.

This study randomly allocated groups through a randomization system, and entered the following treatment groups at a ratio of 1:1: (1) Experimental group: mfolfox6 and hlx04 regimen induction therapy followed by slulimab treatment (36 cases); (2) Control group Group: mfolfox6 and hlx04 regimen treatment (36 cases).

DETAILED DESCRIPTION:
Colorectal Cancer (CRC) is a common malignant tumor. Its incidence ranks third and second among men and women respectively, and its mortality rate ranks third. Data from the World Health Organization's International Agency for Research on Cancer (IARC) in 2020 show that more than 930,000 patients died due to CRC. Since 2000, the incidence and mortality of colorectal cancer have been steadily increasing in China. The National Cancer Center of China (NCC) reported that there were approximately 408,000 new cases of CRC in China in 2016, and approximately 196,000 deaths. Most of the patients are in the mid-to-late stage when diagnosed, and about 35% of them are in the advanced stage. They have no chance of radical surgery and can only receive palliative care.

In the early days when leucovorin (LV) and 5-fluorouracil (5-FU) were used as the main treatment options for patients with metastatic colorectal cancer (mCRC), the efficacy was poor, and the median overall survival (OS) of patients was only for 8-12 months. Since the introduction of effective cytotoxic drugs such as irinotecan and oxaliplatin in 2000, the combination regimens FOLFOX (5-FU/LV + oxaliplatin) and FOLFIRI (5-FU/LV + irinotecan) have become first-line systemic Standard protocol in treatment. The use of biologics targeting key pathways in the development and progression of mCRC, such as epidermal growth factor receptor (EGFR) and vascular endothelial growth factor (VEGF)-related pathways, further extends the survival of mCRC patients.

In the latest version of CSCO colorectal cancer diagnosis and treatment guidelines, the main recommended first-line treatments are FOLFOX/FOLFIRI±bevacizumab or cetuximab (both RAS and BRAF are wild-type), FOLFOX/FOLFIRI±bevacizumab (RAS or BRAF mutant).

PD-1 plays an important role in suppressing immune responses and promoting immune tolerance by inhibiting the activity of T cells, allowing cancer cells to evade immune surveillance. Cells in the tumor microenvironment often express PD-1 and PD-L1. Consistent with the inducible expression of PD-L1 by tumor cells, activated CD8+ effector T cells often express PD-1, indicating that tumor cells are resistant to adaptive immune responses. PD-L1 has been found to be expressed in many types of cancer, including melanoma, lung cancer, urothelial cancer, and hepatocellular carcinoma. Its expression can also be induced by various factors such as radiation, which helps cancer cells evade immune regulation. Blocking the PD-1/PD-L1 interaction has been shown to treat a variety of cancers. Clinical studies have proven that anti-PD-1 and anti-PD-L1 monoclonal antibodies can induce long-lasting anti-tumor activity against a variety of tumors. Anti-PD-1 monoclonal antibodies have been approved for the treatment of melanoma, non-small cell lung cancer, small cell lung cancer, head and neck squamous cell carcinoma, urothelial carcinoma, entities with high microsatellite instability or mismatch repair deficiency and colorectal cancer, gastric cancer, esophageal cancer, cervical cancer, hepatocellular carcinoma (HCC), Merkel cell carcinoma (MCC), renal cell carcinoma, endometrial cancer, bladder cancer, primary mediastinal large B-cell lymphoma ( PMBCL) and classic Hodgkin lymphoma. A large number of clinical studies of anti-PD-1 antibodies are currently underway, some as monotherapy and some in combination with multiple drugs.

This study is an open-label, single-arm, phase II clinical trial. The study inclusion criteria are patients with unresectable mCRC aged 18-75 years old and histologically confirmed by multidisciplinary treatment (MDT). The patients have RAS gene mutations and are confirmed to be MSS. state. All patients received treatment with sintilimab combined with CapeOx and bevacizumab. After the disease achieved complete response (CR)/partial response (PR)/stable disease (SD), maintenance treatment was performed. The main purpose of the study Endpoints include objective response rate (ORR) as assessed by RECIST v1.1 and adverse events as assessed by CTCAE v5.0. The secondary endpoint is progression-free survival (PFS).

This study mainly aims to explore the effectiveness of chemotherapy and bevacizumab induction therapy combined with PD-1 monoclonal antibody in the first-line treatment of MSS-type initial unresectable metastatic colorectal cancer. The second is its safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteered to participate in the study, signed the informed consent form, and had good compliance.
2. Age: 18-75 years old (including 18 years old and 75 years old).
3. Body weight of 40kg.
4. Metastatic colorectal cancer confirmed by histology and / or cytology and initially unresectable.
5. MSS type or pMMR.
6. Patients are required to have at least one measurable lesion (RECIST 1.1).
7. ECOG physical strength status: 0-1 point.
8. Expected survival of 12 weeks.
9. Blood test (no transfusion within 14 days, no correction with granulocyte colony stimulating factor or other hematopoietic stimulating factor within 7 days before the laboratory test)

   1. Absolute neutrophil value of 1.5109/ L, platelet 1010109/ L, hemoglobin concentration of 9 g/dL);
   2. Liver function test (bilirubin 1.5 ULN; aspartate aminase and glutamate aminase 2.5 ULN, AST and ALT 5 ULN);
   3. Renal function (serum creatinine 1.5 ULN or creatinine clearance (CCr) 60 mL/min);
   4. Coagulation (international normalized ratio (INR) 1.5 ULN, prothrombin time (PT) and activated partial thromboplastin time (APTT) 1.5 ULN);
   5. Thyroid function, upper limit of normal (TSH); if abnormal, FT3 and FT4 levels should be examined, normal FT3 and FT4 levels can be included.
10. Women of childbearing age must have a negative serum pregnancy test within 14 days before treatment and be willing to use medically approved effective contraception (e. g., IU, contraceptives or condoms) during 3 months after the study and the last study drug; surgical sterilization for male subjects with a woman of childbearing age, or effective contraception is recommended during the study and 3 months after the last study dose.

Exclusion Criteria:

1. Have received the following treatments within the first 4 weeks of treatment: tumor radiotherapy, surgery, chemotherapy, immune or molecular targeted therapy, and other clinical study drugs.
2. Active autoimmune diseases requiring systemic treatment (i. e., corticosteroids or immunosuppressive agents) have occurred in the past 2 years. Alternative therapies (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are not considered systemic treatment.
3. Diagnosis with immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first treatment. A physiological dose of corticosteroids may be approved after consultation with the investigator.
4. Previous small molecule targeted drug therapy, such as fuquintinib, etc.
5. Previous treatment with an oxaliplatin-based chemotherapy regimen.
6. Symptomatic brain or meningeal metastases.
7. Metastatic colorectal cancer with either MSI-H or dMMR.
8. Severe infection (e. g. intravenous infusion of antibiotics, antifungals or antiviral drugs), or unexplained fever> 38.5℃ during screening / first dose.
9. Hypertension that is not well controlled with antihypertensive medication (systolic 140 mmHg or diastolic 90 mmHg).
10. Significant clinical bleeding symptoms or significant bleeding tendency (bleeding> 30 mL, hematemesis, black feces, stool within 3 months), hemoptysis (> 5 mL of fresh blood within 4 weeks); or venous / venous thrombosis events within 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism; or long-term anticoagulation with Chinese standard or heparin, or long-term antiplatelet therapy (aspirin 300 mg / day or clopidogrel 75 mg / day).
11. During screening, the tumor was found to invade large vascular structures, such as pulmonary artery, superior vena cava vein or inferior vena cava vein, which was judged to be at risk of large bleeding by the investigators.
12. Active heart disease, including myocardial infarction, severe / unstable angina, within 6 months before treatment. Echocardiography showed a left ventricular ejection fraction of <50%, and the arrhythmia was poorly controlled.
13. Other malignancies within or during the previous 5 years (except for cured skin basal cell carcinoma and carcinoma of the cervix in situ).
14. Known allergy to the study drug or any of its excipients.
15. Active or uncontrolled serious infection; A)known human immunodeficiency virus (HIV) infection; B) known history of clinically significant liver disease, including: viral hepatitis [known hepatitis B virus (HBV) carriers must exclude active HBV infection, namely HBV DNA positive (> 1104 copies / mL or> 2000 IU / mL); known hepatitis C virus infection (HCV) and HCV RNA positive (> 1103 copies / mL)], or other hepatitis, cirrhosis;
16. Any other disease, clinically significant metabolic abnormalities abnormal physical examination or laboratory abnormalities, according to the investigator, there is reason to suspect a disease or state is not suitable for the study drug (such as seizures and need treatment), or will affect the interpretation of the results, or make the patient in a high risk situation.
17. Routine urine indicates urine protein 2 +, and 24-hour urine protein quantification> 1.0g.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival（PFS） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  The time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
objective response rate(ORR) | through study completion, an average of 1 year
  It refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time
disease control rate(DCR) | through study completion, an average of 1 year
  Refers to the proportion of patients with best overall assessment of complete response, partial response, or stable disease.
overall survival(OS) | 5 years
  Overall survival (os) is defined as the date from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shao hospital, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No